CLINICAL TRIAL: NCT06487234
Title: Determining the Physiological Mechanism Behind Acute ObeEnd Device Exposure on Factors Regulating Appetite
Brief Title: Effect of Acute ObeEnd Exposure on Factors Regulating Appetite
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 30015229
Record Dates: First submitted 2024-05-30; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-05

CONDITIONS: Obesity
Keywords: Acupuncture; Wearable wellness device
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional band (Active Comparator)
  Interventions: Device: Functional band
- Nonfunctional band (Placebo Comparator)
  Interventions: Device: Placebo band

INTERVENTIONS:
Device: Functional band — Participants will wear the functional band for 1-hour electroacupuncture stimulation
  Arms: Functional band
Device: Placebo band — Participants will wear the nonfunctioning band for 1-hour with no electroacupuncture stimulation
  Arms: Nonfunctional band

SUMMARY:
n Canada, over 60% of adults are classified as overweight and obese resulting in a public health crisis including increasing health care costs and negatively impacting the well-being of many Canadians. To overcome these barriers, the ObeEnd device, manufactured by WAT Medical Enterprise, is a new and innovative wellness technology that uses electrical pulses to stimulate acupressure point PC6 to help control appetite. PC6 stimulation could potentially modulate appetite and restore gastric dysfunction, which are important factors that contribute to obesity. If PC6 electrostimulation facilitates the normalization of appetite and restoration of gastric dysfunction in those with obesity, then the device could be a potentially helpful aid to weight loss.

To measure the change of appetite hormones and enzymes related to appetite regulation after using the ObeEnd device. The investigators hypothesize that, compared to placebo, acute electrostimulation of PC6 an acupuncture spot on the wrist for a 1 hour period will result in changes in enterogastric hormones in a direction that decreases appetite. This study will provide the first evidence of the acute effects of electrostimulation at PC6 on factors affecting body weight regulation providing insight into the utility of the ObeEnd device for weight control.

ELIGIBILITY:
Inclusion Criteria:

* People with obesity (BMI>30kg/m2)
* Generally healthy
* Premenopausal females

Exclusion Criteria:

* Past (<1 year) or present use of nicotine products
* History of chronic disease or metabolic conditions
* Females who are pregnant, less than 6 months postpartum, or breastfeeding
* Diagnosed hepatic disease, renal impairment, uncontrolled hypothyroidism
* Use of any medications that may affect study outcomes (e.g. hormone replacement therapy)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-05 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Appetite assessment | Baseline to 4 hours
  Perceived appetite as reported based on the Visual Analog Scale after a standardized mixed meal. Appetite will be assessed every 30 minutes over a 2 hour period post meal consumption, at 30, 60, 90 and 120 minutes. The Visual Analog Scale is a measure of appetite based on a 10 cm line. Participants are asked a question on how they feel about a specific aspect of appetite (e.g. hunger). Participants then place a mark on the line. A mark closer to the left indicates fullness and satiation and a mark closer to the right indicates hunger.
Blood Hormones | Baseline to 4 hours
  Fasting blood hormone levels will be measured prior to stimulation, and every 30 minutes over a 2 hour period post meal consumption, (at 30, 60, 90 and 120 minutes). Blood hormones involved in appetite and motility such as ghrelin, glucagon-like peptide 1, motilin, and pepsinogen-1 will be measured via ELISA.

SECONDARY OUTCOMES:
Blood Pressure | Baseline to after stimulation, on average 1 hour
  Blood pressure will be measured (mmHg)
Heart rate | Baseline to after stimulation, on average 1 hour
  Heart rate will be measured (beats per minute)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Santosa, PhD, RD, Principal Investigator — Concordia University, Montreal
Locations (1):
- Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
On request and approval by ethics
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available after the study results have been accepted for publication. The data will be available for 5 y.
Access Criteria: On request with ethics approval.